CLINICAL TRIAL: NCT05348408
Title: Efficacy of Ultra-sound Guided Peri-neural Platelet Rich Plasma Injection in Treatment of Chemotherapy Induced Peripheral Neuropathy: Randomized Controlled Trial.
Brief Title: Efficacy of Peri-neural Platelet Rich Plasma Injection in Treatment of Chemotherapy Induced Peripheral Neuropathy.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Nayira Mahmoud El-Husseini, Assistant lecturer of Anesthesia, ICU and pain releis, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 573
Record Dates: First submitted 2022-04-13; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- platelet rich plasma (Active Comparator): patients will be injected perineural platelet rich plasmawith 1.5 to 3 ml around each affected nerve
  Interventions: Drug: platelet rich plasma
- contact group (Sham Comparator): only medical treatment in form of opioid and NSAIDs will be used
  Interventions: Drug: platelet rich plasma

INTERVENTIONS:
Drug: platelet rich plasma — perineural PRP injection under ultrasound guidance in addition to medical treatment
  Other Names: medical treatment

SUMMARY:
This study aims to show the efficacy and safety of ultra-sound guided peri-neural platelet rich injection in treatment of chemotherapy induced peripheral neuropathy.

DETAILED DESCRIPTION:
This study is prospective, randomized, assessor blinded controlled trial. It is aims to study the effect of perineural platelet rich plasma injection in cancer patients with prepheral neuropathy despite of stoppage chemotherapy for 6 months and usage of medical treatment.

Ultrasound-guided PRP injection will be performed after preparation of plasma obtained from the patient by using 10-19 MHz high frequency linear transducer to scan the superficial nerves.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients with peripheral neuropathy confirmed by clinical evaluation and nerve conduction study despite of medical treatment

Exclusion Criteria: patients with:

* Foot ulcers and / or amputation.
* Peripheral vascular disease.
* Uncontrolled diabetes
* Vertebral pathologies.
* Connective tissue diseases.
* Thyriod disorders, significant renal or hepatic dysfunction.
* Platelet dysfunction syndrome, critical thrombocytopenia.
* Septicemia and local infection at the site of the procedure.
* Systemic corticosteriod adminstiration or local injection at the suspected treatment site within the last month.
* Recent fever or illness.
* Hemoglobin level less than 10 g/dl, platelet count less than 105-109/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change in severity of pain after injection | baseline, 15 days, 1 month, 2 months, 3 months
  Change in severity of pain after prp injection wii be assessed using a 10-cm Visual Analog Scale (0 = no pain and 10 =worst imaginable pain

SECONDARY OUTCOMES:
total neuropathy score | baseline, 15 days, 1 month, 2 months, 3 months
  used by non neurologists in oncology practice setting, includes items that quantify pinprick sensation, tuning fork-based vibration thershold, deep tendon reflex, strength. score range 0-28
The functional Asseeement of Cancer Therapy/Gynecological Cancer Group-Neurotoxicity questionnaire (FACT/GOG-Ntx) | baseline, 15 days, 1 month, 2 months, 3 months
  a 27 questionnaire that measure health related quality of life in patients with cancer ad chronic illnesses
Nerve conduction study | baseline, 3 months
  To measure how fast the electrical impulses moves through the nerve.
A 7- point Likert like verbal rating scale | baseline, 15 days, 1 month, 2 months, 3 months
  extremely dissatisfied = 1, dissatisfied = 2, somewhat dissatisfied = 3, undecided = 4, somewhat satisfied = 5, satisfied = 6 and extremely satisfied = 7

IPD SHARING:
Plan to Share IPD: No